CLINICAL TRIAL: NCT02216474
Title: Brain Stimulation in Movement Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birmingham and Solihull Mental Health NHS Foundation Trust (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 14/WM/0119-NRR1301
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Huntington's Disease; Tourette Syndrome
MeSH Terms: conditions — Huntington Disease; Tourette Syndrome | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham transcranial direct current stimulation (frontal cortex) (Sham Comparator): Transcranial direct current stimulation will be ramped up over 60 seconds and then ramped down gradually to encourage blinding to condition.
  Interventions: Other: Transcranial direct current stimulation
- Anodal transcranial DC stimulation (frontal cortex) (Experimental): Anodal transcranial direct current stimulation to prefrontal cortex for approximately 15 minutes plus ramp up and down time
  Interventions: Other: Transcranial direct current stimulation

INTERVENTIONS:
Other: Transcranial direct current stimulation

SUMMARY:
Brain stimulation in movement disorders

This trial will explore the effects of very gentle electrical stimulation of the brain in patients with movement disorders. Other studies have already been carried out and have shown that brain stimulation may help to improve mental abilities and the symptoms of conditions such as depression and stroke. The investigators will show whether this method can help with symptoms such as memory and concentration problems in patients with movement disorder who have mild to moderate problems with these mental abilities. The investigators will also look at the effects of brain stimulation on movement symptoms and mood. These people will be compared to healthy people to help us understand whether brain stimulation works differently in healthy people and people with brain disorders.

This trial is being carried out at one centre in Birmingham. It is scheduled to begin in September 2014 and will last for up to five years. As the study commences it is being funded by Birmingham and Solihull Mental Health Foundation Trust and University of Birmingham. The investigators plan to recruit up to a maximum of 200 individuals in this study.

DETAILED DESCRIPTION:
The procedure does not involve any surgery or hair removal. We simply put a small amount of electrode gel on your head and then hold two electrodes on the top of your head for a short period of time (15-20 minutes) while they generate a small electrical current. It is quite common for participants to feel a tingling or an itch near where the electrode is applied, but if so, this usually wears off within a few minutes. Previous research has shown this method can occasionally lead to mild side-effects (e.g. headache, nausea, fatigue, exacerbation of scalp skin conditions). However, there are no known harmful long term effects. The positive benefits of brain stimulation can include improving the functioning of the brain for a short while after the stimulation session, in a way that may help with things like memory problems. Some people may not notice any change, but an improvement may still be detected using tests of complex mental skills including memory tasks. It is also possible that mood symptoms (e.g. depressive thoughts) could improve. The study will explore these possibilities. Looking at whether brain stimulation can help with health symptoms can help us develop new treatments.

This trial will include patients with two different movement disorders: Tourette syndrome and Huntington's disease. In both of these conditions, changes deep within the brain can have a knock on effect on higher brain areas important for complex mental abilities, as well as brain areas involved in movement control. Participants will be male and female adults (aged 18-65). Patients will have either Tourette syndrome (as diagnosed according to current medical criteria) or Huntington's disease (diagnosed by a genetic test). Patients will have few (if any) signs of additional medical conditions. Healthy controls (who will be compared to patients) will have no current significant medical or psychiatric diagnoses, history of drug use or brain injury.

There will be least two separate appointments for you to attend the study center. We will first assess your mental abilities (e.g. memory, attention) and interview you about current mood or medical symptoms. Brain stimulation will be given to slightly different areas of the outer part of the brain, near the top and front of the head, for each patient group. You may be asked to take part in the trial where there is a no-treatment placebo condition, where the procedure will feel similar to real brain stimulation, but real brain stimulation will not take place. If you receive the placebo condition you will also receive real stimulation, but you will not know which condition is which. This means the effects of expectations are less likely to influence the results. After brain stimulation we will take measures of mental abilities, and compare them to measures taken before brain stimulation, to show whether brain stimulation has had a greater effect on mental abilities than expected by chance.

You may be asked to complete a simple task (e.g. remembering numbers) while having the brain stimulation, as it has been suggested that this could make the effects of stimulation more effective in improving mental skills. As the trial continues, some participants will be invited to have repeated sessions of stimulation over a few days (e.g. three appointments over three days in a row) to look at whether this could make the effects last longer. We will record the effects of brain stimulation on participant's mental skills, movement symptoms and mood, as well as any side effects. We will collect data about your symptoms and health conditions in order to look for relationships between these factors and the effects of brain stimulation. Finally, you may be asked to have a brain scan straight after receiving brain stimulation, so we can look for any changes in brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have either Tourette syndrome (TS) diagnosed according to Diagnostic and Statistical Manual of Mental Disorders criteria or Huntington's disease (HD) diagnosed genetically
* Controls will be generally healthy individuals not taking any psychoactive medications and without diagnosed psychiatric or serious medical conditions (e.g. history of seizures, heart disease, head injury)
* 18-65 years of age for TS; 40-65 years of age for HD; 18-65 for controls
* English as a first language

Exclusion Criteria:

* No current significant co-morbid psychiatric disorder (e.g. learning disability, schizophrenia) or medical condition which may contraindicate brain stimulation or magnetic resonance imaging (e.g. epilepsy, chronic heart disease, scalp skin conditions, metal skull implants). Mild symptoms of obsessive compulsive disorder, attention deficit hyperactivity disorder and/or mood disorders will be accepted as these are very common
* No contraindications to MRI scanning (if they will be scanned) such as metal in the body, claustrophobia or seizure history
* No complex medication regimes (e.g. combinations of multiple dopaminergic drugs plus selective serotonin reuptake inhibitors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-09; Primary Completion 2018-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function (working memory, response inhibition) | From baseline to five minutes after brain stimulation and from baseline to two weeks after stimulation (follow-up)

SECONDARY OUTCOMES:
Change in motor symptom severity (tics/chorea) | From baseline to five minutes after brain stimulation and from baseline to two weeks after stimulation (follow-up)
Mood change (anxiety and depression questionnaire scores) | From baseline to five minutes after brain stimulation and from baseline to two weeks after stimulation (follow-up)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuropsychiatry, BSMHFT The Barberry, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Eddy CM, Shapiro K, Clouter A, Hansen PC, Rickards HE. Transcranial direct current stimulation can enhance working memory in Huntington's disease. Prog Neuropsychopharmacol Biol Psychiatry. 2017 Jul 3;77:75-82. doi: 10.1016/j.pnpbp.2017.04.002. Epub 2017 Apr 5. PMID 28390970